CLINICAL TRIAL: NCT05157412
Title: Role of Doxycycline in the Management of Patients With Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Role of Doxycycline in Chronic Rhinosinusitis With Nasal Polyps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Essam Ali AbuElmagd, Residant, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Doxycycline in Nasal Polyps
Record Dates: First submitted 2021-10-25; First posted 2021-12-15 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Nasal Polyps; Chronic Rhinosinusitis With Nasal Polyps
MeSH Terms: conditions — Nasal Polyps | interventions — Doxycycline; Tablets; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Steroids + Doxycycline (Experimental): Systemic Prednisolone in decreasing doses (40 mg/d on days 1-7, 20 mg/d on days 8-14, and 10 mg/d on days 15-21) along with Doxycycline (200 mg as a loading dose on the 1st day, followed by 100 mg once daily one hour before meal as a maintenance dose) for 3 weeks.
  Interventions: Drug: Doxycycline 100 mg Oral Tablet; Drug: Prednisolone 20 mg
- Steroids Only (Active Comparator): Systemic Prednisolone in decreasing doses (40 mg/d on days 1-7, 20 mg/d on days 8-14, and 10 mg/d on days 15-21) for 3 weeks.
  Interventions: Drug: Prednisolone 20 mg

INTERVENTIONS:
Drug: Doxycycline 100 mg Oral Tablet — Oral Doxycycline will be added to prednisolone as a comparison to using prednisolone as a sole therapy for the treatment of nasal polyps associated with chronic rhinosinusitis
  Other Names: doxycycline
  Arms: Steroids + Doxycycline
Drug: Prednisolone 20 mg — Prednisolone will be used in both arms as a sole therapy in one and together with doxycycline in the other
  Other Names: prednisolone

SUMMARY:
To evaluate the efficacy of Doxycycline as an adjunct to systemic steroids in the treatment of chronic rhinosinusitis with nasal polyps

DETAILED DESCRIPTION:
Chronic rhinosinusitis with nasal polyps (CRSwNP) is a disease of the nose and paranasal sinuses characterized by mucosal thickening and polyp formation. The prevalence of CRSwNP in the general population ranges between 1 and 4%. It mostly affects adult individuals. The treatment of CRSwNP can include the use of steroids, antibiotics, saline nasal spray, mucolytics, topical/systemic decongestants, topical anticholinergics, anti-leukotrienes or receptor blockers, and antihistamines. Steroids have a multitude of effects, including inhibition of cytokine synthesis, reduction of the number of eosinophils and activated eosinophils, anti-oedema effects and reduction of transudation. Topical corticosteroid therapy is not effective in all patients, leading to the use of systemic glucocorticosteroids and/or sinus surgery to control the disease. As a new approach, antibiotics are being used to treat CRSwNP particularly in patients with disease exacerbated by the Staphylococcus aureus enterotoxin. Antibiotics with anti- inflammatory effects can be used to treat patients with chronic rhinosinusitis without polyps, which might be the precursor to CRSwNP. Long-term treatment with these drugs, in selected cases, may be effective when corticosteroids fail. Doxycycline has dual action: it has well described, broad-spectrum antibacterial activity against S aureus as well as anti-inflammatory properties. It appears to be effective in treatment of several chronic inflammatory airway diseases.

ELIGIBILITY:
Inclusion Criteria:

1- Adult patients (aged 18 and over) with bilateral nasal polyps confirmed by nasal endoscopy and CT scan.

Exclusion Criteria:

1. CRS without nasal polyps.
2. Unilateral nasal polyps.
3. Pregnant and lactating women.
4. Patients younger than 18 years old.
5. Subjects with known allergic reaction to steroids or tetracyclines, hypertension, diabetes (type 1 and 2), glaucoma, tuberculosis, herpes infection are excluded.
6. If any major complications to the drugs in use appeared in process.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Polyp Size Score by Nasal Endoscopy | after 12 weeks from the start of treatment
  Every patient will undergo nasal endoscopy at the initial visit and every follow-up visit using a modified Lildholdt scoring system and given scores from 0 to 4. The total nasal polyp score is the sum of the scores from the right and left nostrils.
  0 = No polyps.
  1. = Small polyps in the middle meatus not reaching below the inferior border of the middle concha.
  2. = Polyps reaching below the lower boarder of the middle turbinate.
  3. = Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle concha.
  4. = Large polyps causing almost complete obstruction of the inferior meatus.
Radiological Evaluation | after 12 weeks from the start of treatment
  Multislice computed tomography scan of the nose and paranasal sinuses will be done before starting the treatment and at the end of the follow-up period (12 weeks) using the Lund-Mackay (LMK) scoring system where each sinus (maxillary, anterior ethmoidal, posterior ethmoidal, frontal, sphenoidal) is scored for opacification (0, no opacity; 1, partial opacity; 2, total opacity), and the osteo-meatal complex is scored 0 (no obstruction) or 2 (obstruction). The unilateral score goes from 0 to 12 whereas the bilateral score goes from 0 to 24

SECONDARY OUTCOMES:
Laboratory Measures | after 12 weeks from the start of treatment
  Complete Blood count specifically the eosinophilic count (both relative and absolute) will be documented at the initial visit and at the end of treatment. Values of each group will be compared to each other.
Symptomatology | after 12 weeks from the start of treatment
  Using a questionnaire, all subjects will be asked to evaluate five symptoms (nasal obstruction, Rhinorrhea, postnasal discharge, hyposmia and facial pain) from 0 to 4.
  0 = no symptoms
  1. = mild symptoms
  2. = moderate symptoms
  3. = severe symptoms
  4. = very severe symptoms (intolerable) This will be assessed at the screening visit and follow-up visits at 3, 8 and 12 weeks as a sum of the five individual symptoms of a total score of 20.

CONTACTS AND LOCATIONS:
Overall Officials: Mai AbuElmagd, Principal Investigator — Assiut University; Hamza El Shafie, Study Director — Assiut University; Aly Ragaie, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Van Zele T, Gevaert P, Holtappels G, Beule A, Wormald PJ, Mayr S, Hens G, Hellings P, Ebbens FA, Fokkens W, Van Cauwenberge P, Bachert C. Oral steroids and doxycycline: two different approaches to treat nasal polyps. J Allergy Clin Immunol. 2010 May;125(5):1069-1076.e4. doi: 10.1016/j.jaci.2010.02.020. PMID 20451040
- [Background] Andrews AE, Bryson JM, Rowe-Jones JM. Site of origin of nasal polyps: relevance to pathogenesis and management. Rhinology. 2005 Sep;43(3):180-4. PMID 16218510
- [Background] Tetik F, Korkut AY, Kaya KS, Ucak I, Celebi I, Coskun BU. Comparison of the Oral Steroids, Macrolides and Combination Therapy in Nasal Polyposis Patients. Sisli Etfal Hastan Tip Bul. 2020 Jun 12;54(2):211-217. doi: 10.14744/SEMB.2018.40316. eCollection 2020. PMID 32617061
- [Background] Stammberger H. Rhinoscopic surgery. In: Settipane GA, Lund VJ, Bernstein JM, Tos M, editor. Nasal polyps: epidemiology, patho- genesis and treatment. Rhode Island: Ocean Side Pub; 1997. p.7-15.
- [Background] Hissaria P, Smith W, Wormald PJ, Taylor J, Vadas M, Gillis D, Kette F. Short course of systemic corticosteroids in sinonasal polyposis: a double-blind, randomized, placebo-controlled trial with evaluation of outcome measures. J Allergy Clin Immunol. 2006 Jul;118(1):128-33. doi: 10.1016/j.jaci.2006.03.012. Epub 2006 May 19. PMID 16815148
- [Background] Van Zele T, Gevaert P, Watelet JB, Claeys G, Holtappels G, Claeys C, van Cauwenberge P, Bachert C. Staphylococcus aureus colonization and IgE antibody formation to enterotoxins is increased in nasal polyposis. J Allergy Clin Immunol. 2004 Oct;114(4):981-3. doi: 10.1016/j.jaci.2004.07.013. No abstract available. PMID 15480349
- [Background] Hashiba M, Baba S. Efficacy of long-term administration of clarithromycin in the treatment of intractable chronic sinusitis. Acta Otolaryngol Suppl. 1996;525:73-8. PMID 8908275
- [Background] Legent F, Bordure P, Beauvillain C, Berche P. A double-blind comparison of ciprofloxacin and amoxycillin/clavulanic acid in the treatment of chronic sinusitis. Chemotherapy. 1994;40 Suppl 1:8-15. doi: 10.1159/000239310. PMID 7805431
- [Background] Subramanian HN, Schechtman KB, Hamilos DL. A retrospective analysis of treatment outcomes and time to relapse after intensive medical treatment for chronic sinusitis. Am J Rhinol. 2002 Nov-Dec;16(6):303-12. PMID 12512904
- [Background] Rempe S, Hayden JM, Robbins RA, Hoyt JC. Tetracyclines and pulmonary inflammation. Endocr Metab Immune Disord Drug Targets. 2007 Dec;7(4):232-6. doi: 10.2174/187153007782794344. PMID 18220943